CLINICAL TRIAL: NCT04205812
Title: A Randomized, Double Blind, Phase 3 Study of Platinum-Based Chemotherapy With or Without INCMGA00012 in First-Line Metastatic Squamous and Nonsquamous Non-Small Cell Lung Cancer (POD1UM-304)
Brief Title: Platinum-Based Chemotherapy With/Without INCMGA00012, an Anti-PD-1 Antibody, in Non-Small Cell Lung Cancer
Acronym: POD1UM-304
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCMGA 0012-304; 2019-003372-39 (EudraCT Number); 2022-501987-16-00 (Registry Identifier: EU CT Number)
Expanded Access: NCT06910137 (Available)
Record Dates: First submitted 2019-12-18; First posted 2019-12-19 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Squamous Non-Small Cell Lung Cancer; Metastatic Nonsquamous Non-Small Cell Lung Cancer
Keywords: Metastatic; non-small cell lung cancer; nonsquamous; squamous; PD-1; PD-L1
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin; Carboplatin; Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- INCMGA00012 + chemotherapy (nonsquamous NSCLC) (Experimental): INCMGA00012 with pemetrexed + cisplatin OR carboplatin followed by INCMGA00012 plus pemetrexed until progression.
  Interventions: Drug: Retifanlimab; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin
- Placebo + chemotherapy (nonsquamous NSCLC) (Active Comparator): Placebo with pemetrexed + cisplatin OR carboplatin followed by placebo plus pemetrexed until progression. Participants assigned to placebo + chemotherapy will have the option of receiving open-label monotherapy INCMGA00012 in a crossover period after documentation of progressive disease.
  Interventions: Drug: Placebo; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin
- INCMGA00012 + chemotherapy (squamous NSCLC) (Experimental): INCMGA00012 with carboplatin + paclitaxel OR nab-paclitaxel followed by INCMGA00012 until progression.
  Interventions: Drug: Retifanlimab; Drug: Carboplatin; Drug: Paclitaxel; Drug: nab-Paclitaxel
- Placebo + chemotherapy (squamous NSCLC) (Active Comparator): Placebo with carboplatin + paclitaxel OR nab-paclitaxel followed by placebo until progression. Participants assigned to placebo + chemotherapy will have the option of receiving open-label monotherapy INCMGA00012 in a crossover period after documentation of progressive disease.
  Interventions: Drug: Placebo; Drug: Carboplatin; Drug: Paclitaxel; Drug: nab-Paclitaxel

INTERVENTIONS:
Drug: Retifanlimab — INCMGA00012 administered intravenously every 3 weeks on Day 1 of each cycle for up to 35 cycles.
  Other Names: INCMGA00012
  Arms: INCMGA00012 + chemotherapy (nonsquamous NSCLC); INCMGA00012 + chemotherapy (squamous NSCLC)
Drug: Placebo — Placebo administered intravenously every 3 weeks on Day 1 of each cycle for up to 35 cycles.
  Arms: Placebo + chemotherapy (nonsquamous NSCLC); Placebo + chemotherapy (squamous NSCLC)
Drug: Pemetrexed — Pemetrexed administered intravenously every 3 weeks on Day 1 of each cycle.
  Arms: INCMGA00012 + chemotherapy (nonsquamous NSCLC); Placebo + chemotherapy (nonsquamous NSCLC)
Drug: Cisplatin — Cisplatin administered intravenously every 3 weeks on Day 1 of each cycle for 4 cycles.
  Arms: INCMGA00012 + chemotherapy (nonsquamous NSCLC); Placebo + chemotherapy (nonsquamous NSCLC)
Drug: Carboplatin — Carboplatin administered intravenously every 3 weeks on Day 1 of each cycle for 4 cycles.
Drug: Paclitaxel — Paclitaxel administered intravenously every 3 weeks on Day 1 of each cycle for 4 cycles.
  Arms: INCMGA00012 + chemotherapy (squamous NSCLC); Placebo + chemotherapy (squamous NSCLC)
Drug: nab-Paclitaxel — nab-Paclitaxel administered intravenously every 3 weeks on Days 1, 8, and 15 of each cycle for 4 cycles.
  Arms: INCMGA00012 + chemotherapy (squamous NSCLC); Placebo + chemotherapy (squamous NSCLC)

SUMMARY:
The purpose of this study is to assess the efficacy and safety of platinum-based chemotherapy with or without INCMGA00012 in participants with metastatic squamous and nonsquamous non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC (either nonsquamous or squamous) that is Stage IV (AJCC v8).
* No prior systemic treatment for the advanced/metastatic NSCLC
* Able to provide a formalin-fixed archival tumor tissue sample during screening, or a fresh tumor biopsy
* Measurable disease per RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of at least 3 months.
* Willingness to avoid pregnancy or fathering children.
* Adequate organ function as indicated by protocol-specified laboratory values. - Has been fully vaccinated against SARS-CoV-2 or is willing and able to be fully vaccinated against SARS-CoV-2 during the study by starting the vaccination process during screening.

Exclusion Criteria:

* Clinically significant cardiac disease within 6 months of start of study treatment.
* Any major surgery within 3 weeks of the first dose of study treatment.
* Thoracic radiation therapy of > 30 Gy within 6 months of the first dose of study treatment.
* History of peripheral neuropathy ≥ Grade 2 CTCAE v5 for participants who may receive cisplatin, paclitaxel, or nab-paclitaxel.
* Untreated central nervous system metastases and/or carcinomatous meningitis.
* Evidence or history of interstitial lung disease or noninfectious pneumonitis that required systemic steroids.
* Active infection requiring systemic therapy or active tuberculosis. Note: If required by country or local regulations to be tested for COVID-19 during screening, a participant should be excluded if they have a positive test result for SARS CoV-2 infection until both the retesting result is negative and clinical recovery is obtained.
* Superficial bladder cancer, squamous cell carcinoma of the skin, in situ cervical cancer, or other in situ cancers.
* Has contraindications to chemotherapy agents used in the study.
* Has an active autoimmune disease that has required systemic treatment in past 2 years.
* Is receiving systemic antibiotics or steroid therapy ≤ 7 days prior to the first dose of study treatment.
* Has received a live vaccine within 30 days before the first dose of study treatment (and until 90 days after last dose of study drug).

Note: While based on approved SARS-CoV-2 vaccines available worldwide, many vaccines are not live (mRNA and adenovirus vaccines do not contain live virus), if a live vaccine against SARS-CoV-2 is the only available option, prior consultation with the medical monitor should be obtained.

• Has known active HBV or HCV (testing must be performed to determine eligibility)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 583 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2026-08-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (139):
- United States (3):
  - Pacific Cancer Medical Center, Anaheim, California
  - Innovative Clinical Research Institute, Whittier, California
  - Reading Hospital and Medical Center, Reading, Pennsylvania
- Brazil (12):
  - Fundacao Pio Xii Hospital de Cancer de Barretos, Barretos
  - Incan - Instituto Do Cancer - Hospital Pompeia, Caxias do Sul
  - Centro Regional Integrado de Oncologia, Fortaleza
  - Oncosite - Centro de Pesquisa Clinica E Oncologia, Ijuí
  - Clinica de Neoplasias Litoral Ltda, Itajaí
  - Hospital Do Cancer de Londrina, Londrina
  - Instituto Mederi de Pesquisa E Saude, Passo Fundo
  - Hgb - Hospital Giovanni Battista - Mae de Deus Center, Porto Alegre
  - Inca - Instituto Nacional de Cancer, Rio de Janeiro
  - Sao Camilo Oncologia, S?O Paulo
  - Cepho - Centro de Estudos E Pesquisas de Hematologia E Oncologia, Santo André
  - Fundacao Faculdade Regional de Medicina de Sao Jose Do Rio Preto, São José
- Bulgaria (6):
  - Mc Women'S Health-Nadezhda Eood, Sofia
  - Acibadem Cityclinica Mhat Tokuda, Sofia
  - Umhat Sv. Ivan Rilski Ead, Sofia
  - Mhat Serdika Eood, Sofia
  - Multiprofile Hospital For Active Treatment Central Onco Hospital Ood, Sofia
  - Shatod Dr Marko Marko - Varna Ltd, Varna
- China (19):
  - Hunan Cancer Hospital, Changsha
  - The First Affiliated Hospital Sun Yat-Sen University, Guangzhou
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - Hangzhou Cancer Hospital, Hangzhou
  - The First Affiliated Hospital of Zhejiang University, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - University of Science and Technology of China-First Affiliated Hospital (Anhui Provincial Hospital), Hefei
  - The Second Hospital of Anhui Medical University, Hefei
  - Jinan Central Hospital, Jinan
  - Linyi Cancer Hospital, Linyi
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - Shanghai Chest Hospital, Shanghai
  - General Hospital of Tianjin, Tianjing
  - The Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi
  - Henan Cancer Hostipal, Zhengzhou
  - Henan Provincial Peoples Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- Czechia (4):
  - University Hospital Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Olomouc, Olomouc
  - Nemocnice Agel Ostrava - Vitkovice A.S, Ostrava - Vitkovice
  - Fakultni Nemocnice V Motole, Prague
- Georgia (10):
  - High Technology Hospital Medcenter, Batumi
  - Jsc Evex Hospitals, Kutaisi
  - Archangel St. Michael Multi Profile Clinical Hospital, Tbilisi
  - Israel-Georgian Medical Research Clinic Helsicore, Tbilisi
  - New Hospitals, Tbilisi
  - Medulla Chemotherapy and Immunotherapy Clinic, Tbilisi
  - Tbilisi State Medical University First University Clinic, Tbilisi
  - High Technology Medical Center, University Clinic, Tbilisi
  - Institute of Clinical Oncology Ltd, Tbilisi
  - Cancer Research Center Ltd, Tbilisi
- Hungary (2):
  - Orszagos Koranyi Tbc Es Pulmonological Intezet, Budapest
  - Bacs Kiskun Megyei Oktatokorhaz, Kecskemét
- Malaysia (7):
  - Advanced Medical and Dental Institute Husm, Kepala Batas
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Sarawak General Hospital, Kuching
  - Beacon Hospital Sdn Bhd, Petaling Jaya
  - Hospital Pulau Pinang, Pulau Pinang
  - Institut Kanser Negara - National Cancer Institute, Putrajaya
- Philippines (9):
  - Cebu Doctors University Hospital, Cebu City
  - Asian Hospital and Medical Center, City of Muntinlupa
  - Davao Doctors Hospital, Davao City
  - West Visayas State University Medical Center, Iloilo City
  - Makati Medical Center, Makati
  - Makati Medical Center, Makati City
  - Philippine General Hospital, Manila
  - The Medical City, Pasig
  - St. Lukes Medical Center, Quezon City
- Poland (5):
  - Ko-Med Centra Kliniczne Biala Podlaska, Biała Podlaska
  - Przychodnia Lekarska Komed, Konin
  - Centrum Medyczne Plejady, Krakow
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska Sp. Komandytowo-Akcyjna, Lodz
  - Przychodnia Med-Polonia Sp. Z O.O., Poznan
- Romania (6):
  - S.C Oncopremium Team S.R.L, Baia Mare
  - Institutul Oncologic Prof. Dr. Ion Chiricuta Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic Militar de Urgenta Dr. Constantin Papilian Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Constanta, Constanța
  - S C Oncocenter Oncologie Medicala S R L, Timișoara
  - Oncomed Srl, Timișoara
- Russia (9):
  - Sbih of Arkhangelsk Region Arkhangelsk Clinical Oncological Dispensary, Arkhangelsk
  - Rbih Kursk Regional Clinical Oncology Dispensary of Kursk Region Healthcare Committee, Kursk
  - Federal State Institution "Russian Cancer Research Center Named After N.N. Blokhin" Rams, Moscow
  - Llc Tonus, Nizniy Novgorod
  - Sbhi of Novosibirsk Region Novosibirsk Regional Oncological Dispensary, Novosibirsk
  - Bhi of Omsk Region Clinical Oncology Dispensary, Omsk
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - N.N. Petrov Research Institute of Oncology, Saint Petersburg
  - Sbhi Volgograd Regional Onclogy Dispensary, Volgograd
- Serbia (5):
  - Clinical Center of Serbia, Belgrade
  - Clinical Center Bezanijska Kosa, Belgrade
  - Oncomed-System, Belgrade
  - Institute For Pulmonary Diseases of Vojvodina, Kamenitz
  - Clinical Center Kragujevac, Kragujevac
- South Africa (6):
  - Cape Town Oncology Trials (Pty) Ltd, Cape Town
  - Cancercare Rondebosch Oncology Centre, Cape Town
  - Wits Clinical Research, Johannesburg
  - Sandton Oncology Centre, Johannesburg
  - University of Pretoria Oncology Department, Pretoria
  - Mary Potter Oncology Centre, Pretoria
- Turkey (Türkiye) (15):
  - Acibadem Adana Hospital, Adana
  - Adana Sehir Hastanesi, Adana
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Dr. Abdurrahman Yurtaslan Onkology Teaching and Research Hospital, Ankara
  - Memorial Ankara Hospital, Ankara
  - Yildirim Beyazit University Ankara Ataturk Training and Research Hospital, Ankara
  - Memorial Antalya Hastanesi, Antalya
  - Trakya Universitesi Tip Fakultesi, Edirne
  - Gaziantep University Gaziantep Oncology Hospital, Gaziantep
  - Istanbul University Cerrahpasa - Cerrahpasa Medical Faculty, Istanbul
  - Bakirkoy Dr Sadi Konuk Teaching and Research Hospital, Istanbul
  - Medipol University Medical Faculty, Istanbul
  - Izmir Medicalpark Hospital, Izmir
  - Necmettin Erbakan Universitesi Meram Tip Fakultesi Hastanesi, Konya
  - Inonu Universitesi Turgut Ozal Tip Merkezi, Malatya
- Ukraine (14):
  - Multifield Clinical Hospital No 4, Dnipro
  - Ci Carpathian Clinical Oncological Center, Ivano-Frankivsk
  - Communal Non-Profit Enterprise Regional Center of Oncology, Kharkiv
  - V.T.Zaycev Institute of General and Urgent Surgery of National Academy Medical Sciences of Ukraine, Kharkiv
  - Kherson Regional Oncologic Dispensary, Kherson
  - Pp Ppc Acinus Medical and Diagnostic Centre, Kropyvnytskyi
  - Mi Kryviy Rih Center of Dnipropetrovsk Regional Council, Kryvyi Rih
  - Kyiv City Clinical Oncological Center, Kyiv
  - Medical Center Asklepion Llc, Kyiv
  - Ci of Krc Kyiv Regional Oncologic Dispensary, Kyiv
  - Volyn Regional Oncological Dispensary, Lutsk
  - Rmi Sumy Regional Clinical Oncology Dispensary, Sumy
  - Cne Ccch of Uzh Cc Oncological Center, Uzhhorod
  - Medical Center Oncolife Llc, Zaporizhzhia
- Vietnam (7):
  - Can Tho Oncology Hospital, Can Tho
  - 103 Military Hospital, Hanoi
  - Bach Mai Hospital, Hanoi
  - Hanoi Oncology Hospital, Hanoi
  - National Cancer Hospital, Hanoi
  - National Lung Hospital, Hanoi
  - Hcmc Oncology Hospital, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- [Derived] Lu S, Vynnychenko O, Kulyaba Y, Kuchava V, Ibrahim A, Moiseenko F, Arslan C, Nguyen DT, Petrovic M, Cicin I, Bibichadze K, Cil T, Shi J, Olmez OF, Gogishvili M, Artac M, Nguyen HG, Cornfeld M, Tian C, Munteanu MC, Sette CVM, Bondarenko I; POD1UM-304 Study Team. Retifanlimab versus placebo in combination with platinum-based chemotherapy in patients with first-line non-squamous or squamous metastatic non-small-cell lung cancer (POD1UM-304): a phase 3, multiregional, placebo-controlled, double-blind, randomised study. Lancet Respir Med. 2025 Dec;13(12):1096-1107. doi: 10.1016/S2213-2600(25)00209-7. Epub 2025 Sep 19. PMID 40983066

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted in Bulgaria, Brazil, China, Czech Republic, Georgia, Malaysia, Philippines, Poland, Romania, Russia, Serbia, Turkey, Ukraine, United States, Vietnam, and South Africa. Data collected through 15 December 2023 have been included in this results summary.
Groups:
- Placebo + Chemotherapy: Participants received placebo intravenously (IV) every 3 weeks (Q3W) along with a standard-of-care chemotherapy regimen in the randomized treatment period. Participants with nonsquamous non-small cell lung cancer (NSCLC) received placebo IV (on Day 1 [D1]) Q3W with pemetrexed 500 milligrams per meters squared (mg/m^2) + either cisplatin 75 mg/m^2 (on D1) Q3W or carboplatin AUC 5 (on D1) Q3W for 4 cycles (21-day cycles) followed by placebo IV Q3W + pemetrexed 500 mg/m^2 Q3W until progression. Participants with squamous NSCLC received placebo IV (on D1) Q3W with carboplatin AUC 6 (D1) + either paclitaxel 200 mg/m^2 (on D1) or nab-paclitaxel 100 mg/m^2 (on D1, D8, D15) Q3W for 4 cycles followed by placebo IV Q3W until progression. Treatment could continue for up to 2 years until unacceptable toxicity, disease progression, investigator's decision, pregnancy, withdrawal of consent, or study termination. Participants who experienced progressive disease per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) verified by blinded independent central review (BICR) had the opportunity to receive retifanlimab 375 mg IV Q3W for up to approximately 2 years (or up to 35 cycles [21-day cycles]) in the optional monotherapy treatment period.
- Retifanlimab + Chemotherapy: Participants received retifanlimab 375 mg IV Q3W along with a standard-of-care platinum-based chemotherapy regimen in the randomized treatment period. Participants with nonsquamous NSCLC received retifanlimab 375 mg IV (on D1) Q3W with pemetrexed 500 mg/m^2 + either cisplatin 75 mg/m^2 (on D1) Q3W or carboplatin AUC 5 (on D1) Q3W for 4 cycles (21-day cycles) followed by retifanlimab 375 mg IV Q3W + pemetrexed 500 mg/m^2 Q3W until progression. Participants with squamous NSCLC received retifanlimab 375 mg IV (on D1) Q3W with carboplatin AUC 6 (D1) + either paclitaxel 200 mg/m^2 (on D1) or nab-paclitaxel 100 mg/m^2 (on D1, D8, D15) Q3W for 4 cycles followed by retifanlimab 375 mg IV Q3W until progression. Treatment could continue for up to 2 years until unacceptable toxicity, disease progression, investigator's decision, pregnancy, withdrawal of consent, or study termination.
Period: Randomized Treatment Period
Arm/Group | Placebo + Chemotherapy | Retifanlimab + Chemotherapy
Started | 192 | 391
Completed | 59 | 0
Not Completed | 133 | 391
Not completed — Ongoing | 28 | 138
Not completed — Death | 94 | 226
Not completed — Lost to Follow-up | 5 | 11
Not completed — Physician Decision | 1 | 4
Not completed — Withdrawal by Subject | 4 | 11
Not completed — Progressive Disease | 0 | 1
Not completed — Met Exclusion Criteria | 1 | 0
Period: Monotherapy Treatment Period
Arm/Group | Placebo + Chemotherapy | Retifanlimab + Chemotherapy
Started | 59 | 0
Completed | 0 | 0
Not Completed | 59 | 0
Not completed — Ongoing | 17 | 0
Not completed — Death | 39 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Chemotherapy | Retifanlimab + Chemotherapy | Total
Number analyzed (Participants) | 192 | 391 | 583
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (8.34) | 62.8 (8.44) | 62.8 (8.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 73 | 116
  Male | 149 | 318 | 467
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 15 | 22
  Not Hispanic or Latino | 184 | 375 | 559
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 127 | 260 | 387
  Black/African-American | 1 | 1 | 2
  Black/White biracial | 2 | 2 | 4
  Asian | 62 | 127 | 189
  Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was defined as the time between the date of randomization and the date of death due to any cause.
Time Frame: up to 39.1 months
Population: Median survival time in months was estimated using the Kaplan-Meier method. The confidence interval for median survival time was calculated using the method of Brookmeyer and Crowley. Full Analysis Set: all participants to whom study treatment had been assigned by randomization. Participants were analyzed according to the treatment and strata they had been assigned to during the randomization procedure.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Placebo + Chemotherapy: Participants received placebo intravenously (IV) every 3 weeks (Q3W) along with a standard-of-care chemotherapy regimen in the randomized treatment period. Participants with nonsquamous non-small cell lung cancer (NSCLC) received placebo IV (on Day 1 [D1]) Q3W with pemetrexed 500 milligrams per meters squared (mg/m^2) + either cisplatin 75 mg/m^2 (on D1) Q3W or carboplatin AUC 5 (on D1) Q3W for 4 cycles (21-day cycles) followed by placebo IV Q3W + pemetrexed 500 mg/m^2 Q3W until progression. Participants with squamous NSCLC received placebo IV (on D1) Q3W with carboplatin AUC 6 (D1) + either paclitaxel 200 mg/m^2 (on D1) or nab-paclitaxel 100 mg/m^2 (on D1, D8, D15) Q3W for 4 cycles followed by placebo IV Q3W until progression. Treatment could continue for up to 2 years until unacceptable toxicity, disease progression, investigator's decision, pregnancy, withdrawal of consent, or study termination.
Arm/Group | Placebo + Chemotherapy | Retifanlimab + Chemotherapy
Number analyzed (Participants) | 192 | 391
months | 13.4 [11.0 to 16.7] | 18.1 [16.2 to 21.0]
Statistical Analysis 1: Comparison: Placebo + Chemotherapy vs Retifanlimab + Chemotherapy; Test type: Superiority; p = 0.0042, Log Rank — The p-value was based on a stratified log-rank test at an overall 1-sided 2.5% level of significance, using O'Brien and Fleming boundary to adjust for alpha spending at interim analysis; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.60 to 0.93] — A stratified Cox regression with Efron's method for tie handling was used to estimate the hazard ratio

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the length of time from the date of randomization until the earliest date of disease progression by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1), as determined by blinded independent central review (BICR), or death due to any cause, if occurring sooner than progression.
Time Frame: up to 35.8 months
Population: Full Analysis Set. Median PFS time was estimated using the Kaplan-Meier method. The confidence interval for median PFS time was calculated using the method of Brookmeyer and Crowley.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Chemotherapy | Retifanlimab + Chemotherapy
Number analyzed (Participants) | 192 | 391
months | 5.5 [4.4 to 5.7] | 7.7 [6.9 to 9.0]
Statistical Analysis 1: Comparison: Placebo + Chemotherapy vs Retifanlimab + Chemotherapy; Test type: Superiority; p < 0.0001, Log Rank; The p-value was based on the stratified log-rank test for PFS; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.52 to 0.79] — A stratified Cox regression with Efron's method for tie handling was used to estimate the hazard ratio

3. Secondary Outcome: Objective Response Rate
Description: Objective response rate was defined as the percentage of participants who had a confirmed complete response (CR) or partial response (PR) per RECIST v1.1 based on BICR at any post-Baseline visit until the first progressive disease or new anticancer therapy. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 millimeters (mm). PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions.
Time Frame: up to 35.78 months
Population: Full Analysis Set. Confidence intervals were calculated based on the exact method for binomial distributions.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Chemotherapy | Retifanlimab + Chemotherapy
Number analyzed (Participants) | 192 | 391
percentage of participants | 38.5 [31.6 to 45.8] | 51.7 [46.6 to 56.7]
Statistical Analysis 1: Comparison: Placebo + Chemotherapy vs Retifanlimab + Chemotherapy; Test type: Superiority; p = 0.0012, Cochran-Mantel-Haenszel — The p-value was calculated at the 1-sided 2.5% level from stratified Cochran-Mantel-Haenszel test

4. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from the earliest date of documented response until the earliest date of disease progression or death from any cause, whichever comes first, per RECIST v1.1 based on BICR. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion.
Time Frame: up to 34.3 months
Population: Full Analysis Set. Only those participants with a confirmed response were analyzed. The 95% confidence interval was calculated using the Brookmeyer and Crowley's method and Klein and Moeschberger's method with log-log transformation.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Chemotherapy | Retifanlimab + Chemotherapy
Number analyzed (Participants) | 74 | 202
months | 6.1 [4.2 to 8.3] | 12.7 [9.4 to 15.2]

5. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE) in the Randomized Treatment Period
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. TEAEs were defined as any AEs either reported for the first time or the worsening of pre-existing events after the first dose of retifanlimab/placebo and within 90 days of the last administration of the randomized period. AEs that occurred after new anticancer therapy (including monotherapy treatment) were to be excluded.
Time Frame: up to approximately 39 months
Population: Safety Population: all participants who received at least 1 dose of study treatment. Treatment groups for this population were determined by the actual treatment that the participant received regardless of treatment assignment at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Chemotherapy | Retifanlimab + Chemotherapy
Number analyzed (Participants) | 190 | 389
Participants | 183 | 369

6. Secondary Outcome: Number of Participants Who Discontinued Study Drug Due to TEAEs in the Randomized Treatment Period
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. TEAEs were defined as any AEs either reported for the first time or the worsening of pre-existing events after the first dose of retifanlimab/placebo and within 90 days of the last administration of the randomized period. AEs that occurred after new anticancer therapy (including monotherapy treatment) were to be excluded.
Time Frame: up to approximately 39 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Chemotherapy | Retifanlimab + Chemotherapy
Number analyzed (Participants) | 190 | 389
Participants | 9 | 33

7. Secondary Outcome: Number of Participants With Any TEAE in the Monotherapy Treatment Period
Description: as for outcome 6
Time Frame: up to approximately 27 months
Population: Monotherapy Analysis Set: all participants who were randomized to the placebo group and received at least 1 dose of placebo, who then transitioned and received at least 1 dose of retifanlimab
Measure: Count of Participants; unit: Participants
Groups:
- Retifanlimab Monotherapy: Participants randomized to placebo + platinum-based chemotherapy who experienced progressive disease per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) verified by blinded independent central review (BICR) had the opportunity to receive retifanlimab 375 mg IV Q3W for up to approximately 2 years (or up to 35 cycles [21-day cycles]) in the optional monotherapy treatment period.
Arm/Group | Retifanlimab Monotherapy
Number analyzed (Participants) | 59
Participants | 50

8. Secondary Outcome: Number of Participants Who Discontinued Study Drug Due to TEAEs in the Monotherapy Treatment Period
Description: as for outcome 6
Time Frame: up to approximately 27 months
Population: Monotherapy Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Retifanlimab Monotherapy
Number analyzed (Participants) | 59
Participants | 4

9. Secondary Outcome: Cmax1 of Retifanlimab When Administered With Chemotherapy
Description: Cmax1 was defined as the first-dose maximum serum concentration of retifanlimab.
Time Frame: Cycle 1 Day 1: pre-infusion and immediately after infusion
Population: Pharmacokinetic (PK) Evaluable Population: all participants who received at least 1 dose of retifanlimab and provided at least 1 PK post-dose sample
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams per liter (mg/L)
Arm/Group | Placebo + Chemotherapy | Retifanlimab + Chemotherapy
Number analyzed (Participants) | 0 | 384
milligrams per liter (mg/L) |  | 109 (23.1)

10. Secondary Outcome: AUC1 of Retifanlimab When Administered With Chemotherapy
Description: AUC1 was defined as the first-dose area under the serum concentration versus time curve.
Time Frame: Cycle 1 Day 1: pre-infusion and immediately after infusion
Population: PK Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L x day
Arm/Group | Placebo + Chemotherapy | Retifanlimab + Chemotherapy
Number analyzed (Participants) | 0 | 384
mg/L x day |  | 775 (25.0)

11. Secondary Outcome: Cmaxss of Retifanlimab When Administered With Chemotherapy
Description: Cmaxss was defined as the maximum serum concentration of retifanlimab at steady state.
Time Frame: Cycle 1 Day 1 (C1D1): pre-infusion and immediately after infusion (IAI). C2D1: pre-infusion. C4D1: pre-infusion and IAI. C6D11: pre-infusion. C8D1, and every 4 cycles thereafter: pre-infusion. End of treatment visit and 30-day safety follow-up visit.
Population: PK Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Placebo + Chemotherapy | Retifanlimab + Chemotherapy
Number analyzed (Participants) | 0 | 384
mg/L |  | 109 (23.1)

12. Secondary Outcome: AUCss of Retifanlimab When Administered With Chemotherapy
Description: AUCss was defined as the area under the serum concentration versus time curve at steady state.
Time Frame: as for outcome 11
Population: PK Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L x day
Arm/Group | Placebo + Chemotherapy | Retifanlimab + Chemotherapy
Number analyzed (Participants) | 0 | 384
mg/L x day |  | 791 (23.1)

ADVERSE EVENTS:
Time Frame: up to approximately 3.25 years
Description: All-Cause Mortality was assessed for all randomized participants (Full Analysis Set). Adverse events were assessed for members of the Safety Population (participants who received at least 1 dose of study treatment) and the Monotherapy Analysis Set (participants who were randomized to the placebo group and received at least 1 dose of placebo, who then transitioned and received at least 1 dose of retifanlimab).
Groups:
- Retifanlimab + Chemotherapy: Participants received retifanlimab 375 milligrams (mg) intravenously (IV) every 3 weeks (Q3W) along with a standard-of-care platinum-based chemotherapy regimen in the randomized treatment period. Participants with nonsquamous non-small cell lung cancer (NSCLC) received retifanlimab 375 mg IV (on Day 1 [D1]) Q3W with pemetrexed 500 milligrams per meters squared (mg/m^2) + either cisplatin 75 mg/m^2 (on D1) Q3W or carboplatin AUC 5 (on D1) Q3W for 4 cycles (21-day cycles) followed by retifanlimab 375 mg IV Q3W + pemetrexed 500 mg/m^2 Q3W until progression. Participants with squamous NSCLC received retifanlimab 375 mg IV (on D1) Q3W with carboplatin AUC 6 (D1) + either paclitaxel 200 mg/m^2 (on D1) or nab-paclitaxel 100 mg/m^2 (on D1, D8, D15) Q3W for 4 cycles followed by retifanlimab 375 mg IV Q3W until progression. Treatment could continue for up to 2 years until unacceptable toxicity, disease progression, investigator's decision, pregnancy, withdrawal of consent, or study termination.
- Placebo + Chemotherapy: Participants received placebo IV Q3W along with a standard-of-care chemotherapy regimen in the randomized treatment period. Participants with nonsquamous NSCLC received placebo IV (on D1) Q3W with pemetrexed 500 mg/m^2 + either cisplatin 75 mg/m^2 (on D1) Q3W or carboplatin AUC 5 (on D1) Q3W for 4 cycles (21-day cycles) followed by placebo IV Q3W + pemetrexed 500 mg/m^2 Q3W until progression. Participants with squamous NSCLC received placebo IV (on D1) Q3W with carboplatin AUC 6 (D1) + either paclitaxel 200 mg/m^2 (on D1) or nab-paclitaxel 100 mg/m^2 (on D1, D8, D15) Q3W for 4 cycles followed by placebo IV Q3W until progression. Treatment could continue for up to 2 years until unacceptable toxicity, disease progression, investigator's decision, pregnancy, withdrawal of consent, or study termination.
- Randomized Treatment Period Total: Participants received retifanlimab 375 mg IV Q3W or matching placebo along with a standard-of-care platinum-based chemotherapy regimen in the randomized treatment period.
- Retifanlimab Monotherapy: Participants randomized to placebo plus a platinum-based chemotherapy who experienced progressive disease per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) verified by blinded independent central review (BICR) had the opportunity to receive retifanlimab 375 mg IV Q3W for up to approximately 2 years (or up to 35 cycles [21-day cycles]) in the optional monotherapy treatment period.
Arm/Group | Retifanlimab + Chemotherapy | Placebo + Chemotherapy | Randomized Treatment Period Total | Retifanlimab Monotherapy
All-Cause Mortality (participants affected / at risk) | 234/391 | 140/192 | 374/583 | 42/59
Serious Adverse Events (participants affected / at risk) | 158/389 | 57/190 | 215/579 | 12/59
Other Adverse Events (participants affected / at risk) | 350/389 | 177/190 | 527/579 | 44/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retifanlimab + Chemotherapy (N=389) | Placebo + Chemotherapy (N=190) | Randomized Treatment Period Total (N=579) | Retifanlimab Monotherapy (N=59)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 3 (4) | 7 (8) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 16 (21) | 3 (3) | 19 (24) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Asthenia (General disorders) | 3 (3) | 1 (2) | 4 (5) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 14 (14) | 4 (4) | 18 (18) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 4 (4) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 3 (3) | 1 (1) | 4 (4) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cerebral artery embolism (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 3 (3) | 1 (1) | 4 (4) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 2 (2) | 4 (4) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (11) | 1 (1) | 4 (12) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 1 (3) | 1 (3) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diabetes insipidus (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 0 (0) | 5 (5) | 0 (0)
Dilated cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 9 (9) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 10 (10) | 5 (6) | 15 (16) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 2 (3) | 0 (0) | 2 (3) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 3 (4) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Immune-mediated adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 2 (3) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Lymphangitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (5) | 1 (1) | 6 (6) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Organ failure (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 3 (4) | 0 (0) | 3 (4) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Performance status decreased (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 6 (7) | 2 (2) | 8 (9) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 6 (6) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 25 (30) | 8 (8) | 33 (38) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Post-acute COVID-19 syndrome (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 4 (4) | 15 (15) | 2 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Salmonella bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 4 (6) | 2 (2) | 6 (8) | 0 (0)
Septic shock (Infections and infestations) | 4 (4) | 3 (3) | 7 (7) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 4 (4) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 5 (5) | 0 (0) | 5 (5) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vascular occlusion (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (4) | 1 (1)
White blood cell count decreased (Investigations) | 3 (3) | 1 (1) | 4 (4) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retifanlimab + Chemotherapy (N=389) | Placebo + Chemotherapy (N=190) | Randomized Treatment Period Total (N=579) | Retifanlimab Monotherapy (N=59)
Alanine aminotransferase increased (Investigations) | 72 (125) | 45 (68) | 117 (193) | 9 (15)
Alopecia (Skin and subcutaneous tissue disorders) | 59 (59) | 38 (38) | 97 (97) | 0 (0)
Amylase increased (Investigations) | 20 (30) | 7 (11) | 27 (41) | 2 (3)
Anaemia (Blood and lymphatic system disorders) | 235 (357) | 108 (175) | 343 (532) | 13 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 (33) | 11 (16) | 40 (49) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 68 (124) | 42 (69) | 110 (193) | 14 (22)
Asthenia (General disorders) | 38 (58) | 16 (32) | 54 (90) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 25 (33) | 13 (14) | 38 (47) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 45 (69) | 19 (25) | 64 (94) | 7 (12)
Blood bilirubin increased (Investigations) | 18 (22) | 8 (8) | 26 (30) | 3 (3)
Blood creatine phosphokinase increased (Investigations) | 4 (4) | 1 (1) | 5 (5) | 3 (4)
Blood creatinine increased (Investigations) | 38 (59) | 16 (20) | 54 (79) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 37 (76) | 19 (30) | 56 (106) | 7 (9)
Blood urea increased (Investigations) | 6 (11) | 9 (11) | 15 (22) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 10 (10) | 21 (21) | 1 (1)
COVID-19 (Infections and infestations) | 25 (26) | 8 (8) | 33 (34) | 1 (1)
Constipation (Gastrointestinal disorders) | 56 (83) | 21 (34) | 77 (117) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 55 (73) | 22 (24) | 77 (97) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 88 (115) | 25 (44) | 113 (159) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 49 (66) | 14 (16) | 63 (82) | 4 (5)
Dizziness (Nervous system disorders) | 26 (28) | 12 (12) | 38 (40) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 36 (43) | 15 (15) | 51 (58) | 3 (3)
Electrocardiogram QT prolonged (Investigations) | 6 (16) | 3 (8) | 9 (24) | 3 (4)
Fatigue (General disorders) | 72 (101) | 34 (55) | 106 (156) | 7 (8)
Gamma-glutamyltransferase increased (Investigations) | 30 (36) | 8 (11) | 38 (47) | 4 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 4 (9) | 17 (23) | 3 (3)
Headache (Nervous system disorders) | 28 (42) | 8 (8) | 36 (50) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 50 (98) | 21 (35) | 71 (133) | 6 (11)
Hyperkalaemia (Metabolism and nutrition disorders) | 18 (50) | 9 (12) | 27 (62) | 4 (6)
Hypertension (Vascular disorders) | 21 (32) | 8 (11) | 29 (43) | 1 (2)
Hyperthyroidism (Endocrine disorders) | 35 (44) | 9 (9) | 44 (53) | 4 (5)
Hyperuricaemia (Metabolism and nutrition disorders) | 14 (34) | 8 (13) | 22 (47) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 57 (102) | 29 (39) | 86 (141) | 6 (13)
Hypocalcaemia (Metabolism and nutrition disorders) | 34 (61) | 11 (13) | 45 (74) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 43 (70) | 15 (22) | 58 (92) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 45 (76) | 14 (20) | 59 (96) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 38 (67) | 17 (29) | 55 (96) | 8 (10)
Hypothyroidism (Endocrine disorders) | 31 (45) | 12 (14) | 43 (59) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 35 (56) | 12 (20) | 47 (76) | 0 (0)
Lipase increased (Investigations) | 38 (62) | 9 (11) | 47 (73) | 5 (10)
Lymphocyte count decreased (Investigations) | 41 (124) | 16 (41) | 57 (165) | 3 (8)
Lymphopenia (Blood and lymphatic system disorders) | 21 (36) | 3 (4) | 24 (40) | 0 (0)
Nausea (Gastrointestinal disorders) | 80 (131) | 45 (60) | 125 (191) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 59 (95) | 30 (42) | 89 (137) | 0 (0)
Neutrophil count decreased (Investigations) | 84 (235) | 33 (96) | 117 (331) | 2 (2)
Oedema peripheral (General disorders) | 26 (38) | 10 (10) | 36 (48) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 (35) | 14 (18) | 40 (53) | 2 (2)
Platelet count decreased (Investigations) | 74 (136) | 21 (56) | 95 (192) | 2 (3)
Pneumonia (Infections and infestations) | 32 (38) | 13 (13) | 45 (51) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 29 (44) | 7 (9) | 36 (53) | 4 (6)
Pyrexia (General disorders) | 39 (55) | 12 (15) | 51 (70) | 4 (6)
Rash (Skin and subcutaneous tissue disorders) | 17 (19) | 8 (9) | 25 (28) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 8 (12) | 11 (11) | 19 (23) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 50 (74) | 22 (26) | 72 (100) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 24 (33) | 12 (16) | 36 (49) | 0 (0)
Vomiting (Gastrointestinal disorders) | 38 (52) | 13 (23) | 51 (75) | 3 (6)
Weight decreased (Investigations) | 38 (40) | 18 (19) | 56 (59) | 6 (7)
White blood cell count decreased (Investigations) | 74 (220) | 35 (90) | 109 (310) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT04205812/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/12/NCT04205812/SAP_001.pdf